CLINICAL TRIAL: NCT06681207
Title: An Exploratory Study: The Effects of Cortical Priming on Visuomotor Stepping Learning in Healthy Adults and Persons With Chronic Stroke
Brief Title: Explore the Effects of Cortical Priming on Visuomotor Stepping Learning in Persons With Chronic Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24-0234
Record Dates: First submitted 2024-11-06; First posted 2024-11-08 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Stroke
Keywords: adult; chronic stroke
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Explore the effects of brain stimulation on locomotor skill learning in stroke survivors (Experimental): To explore the trends of locomotor skill learning in three groups: stroke survivors after five sessions of anodal tDCS (a-tDCS, real brain stimulation), stroke survivors after five sessions of sham tDCS (s-tDCS), and stroke survivors with no brain stimulation (control; CON).
  Interventions: Combination Product: anodal transcranial direct current stimulation (a-tDCS)
- determine the effects of a-tDCS on the cortical excitation before and after locomotor learning (Experimental): measure changes in cortical neuronal activation before and after five sessions of locomotor skill training in healthy adults and stroke participants.
  Interventions: Combination Product: anodal transcranial direct current stimulation (a-tDCS)
- To explore improvements in learning capacity between healthy adults and stroke participants. (Experimental): Compare stimulation-induced improvements in learning capacity between three groups: stroke group, healthy young group, and healthy older group.
  Interventions: Combination Product: anodal transcranial direct current stimulation (a-tDCS)
- To explore the trends of functional improvements after five tDCS session in stroke survivors (Experimental): Compare functional improvements (gait performance, balance, motor and cognitive function) between healthy adults and stroke participants after five sessions of brain stimulation.
  Interventions: Combination Product: anodal transcranial direct current stimulation (a-tDCS)

INTERVENTIONS:
Combination Product: anodal transcranial direct current stimulation (a-tDCS) — Stroke participants will be randomly assigned into one of three groups: anodal transcranial direct current stimulation (a-tDCS), sham tDCS (s-tDCS), or control groups (i.e. no brain stimulation). Stroke participants in the first two groups will receive five sessions of the assigned brain stimulation combined with visuomotor stepping training over five consecutive days. Healthy adults will be randomly assignments into a-tDCS or s-tDCS groups.

SUMMARY:
This research study aims to understand the relationship between brain stimulation and leg skill learning in both healthy adults and persons with chronic stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 21 and 90 years
2. Medical history of a unilateral stroke occurring ≥ 6 months prior to enrollment
3. MRI or CT evidence from the imaging report shown that the stroke involves the corticospinal tract
4. Hemiparesis involving the lower extremity (Fulg-Meyer LE motor test)
5. No passive range of motion limitation in bilateral hips and knees
6. Limitation of ankle passive range of motion to 10 degrees of dorsiflexion or less
7. Visual acuity can be corrected by glasses or contact lens to 20/20
8. Able to walk independently with/without assistant devices for 10 meters
9. Able to maintain standing position without any assistance > 30 sec (Short Physical Performance Battery)
10. Evaluation of cognitive status: Mini-mental status examination (MMSE) score ≥ 24

Exclusion Criteria:

1. Pregnant women
2. MRI or CT evidence of involvement of the basal ganglia or cerebellum, evidence of multiple lesions, or evidence of any other brain damage or malignant neoplasm or tumors
3. Have any metal implants, cardiac pacemakers, or history of seizures
4. Ongoing orthopedic or other neuromuscular disorders that will restrict exercise training
5. Any vestibular dysfunction or unstable angina
6. Significant cognitive deficits (inability to follow a 2-step command) or severe receptive or global aphasia*

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-04-23 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in stepping motor control after five sessions of brain stimulation combined with visuomotor stepping learning | Day 1, Day 5, Day 7, Day 30, Day 60, Day 9 post five sessions of brain stimulation combined with visuomotor stepping training
  Stepping motor control will be quantified by the time (seconds) that each participant takes to initiate a forward step onto a visual target displayed on the wall screen.
Mean change from baseline in brain neuronal activations after five sessions of brain stimulation combined with visuomotor stepping learning | Day 1, Day 5, Day 7, Day 30, Day 60, Day 9 post five sessions of brain stimulation combined with visuomotor stepping training
  The neuronal activations will be quantified by peak-to-peak electrical signals detected by surface electromyographic (EMG) electrodes on leg muscles after transcranial magnetic stimulations

SECONDARY OUTCOMES:
Mean change from baseline in lower extremity (LE) motor function after five sessions of brain stimulation combined with visuomotor stepping learning | Day 1, Day 5, Day 7, Day 30, Day 60, Day 9 post five sessions of brain stimulation combined with visuomotor stepping training
  LE motor function will be quantified by Fugl-Meyer LE motor test, Short Physical Performance Battery (SPPB), and gait speed (meters/second) during ground walking tests.
Mean change from baseline in brain neuronal network activations after five sessions of brain stimulation combined with visuomotor stepping learning | Day 1, Day 5, Day 7, Day 30, Day 60, Day 9 post five sessions of brain stimulation combined with visuomotor stepping training
  The neuronal activations will be quantified by oxygen consumption changes locally detected by surface infrared diodes

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Chiao Tseng, PT, PhD, Principal Investigator — University of Texas
Locations (1):
- Physical Therapy, University of Texas Medical Branch, Galveston, Texas, United States